CLINICAL TRIAL: NCT00605397
Title: Pilot Trial of PET Imaging With Cu-64 Labeled Trastuzumab in HER2+ Metastatic Breast Cancer
Brief Title: PET Imaging With Cu-64 Labeled Trastuzumab in HER2+ Metastatic Breast Cancer
Acronym: Cu-64 HER2+
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-134
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Cu-64 LABELED TRASTUZUMAB
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- 1 (Experimental): breast cancer pt receiving trastuzumab therapy will undergo two complete PET studies.
  Interventions: Radiation: PET Imaging With Cu-64 Labeled Trastuzumab
- 2 (Experimental): breast cancer pt receiving trastuzumab therapy will undergo one complete PET studies
  Interventions: Radiation: PET Imaging With Cu-64 Labeled Trastuzumab

INTERVENTIONS:
Radiation: PET Imaging With Cu-64 Labeled Trastuzumab — The first 8 patients enrolled will undergo two complete PET studies, up to 3-6 weeks apart, to assess for reproducibility of measures of tracer uptake into individual organs and known sites of metastatic disease.
  Arms: 1
Radiation: PET Imaging With Cu-64 Labeled Trastuzumab — The remaining 20 patients will undergo one PET study.
  Arms: 2

SUMMARY:
The purpose of this study is to learn more about how a new study agent works inside the body. The study agent is a protein called 64Cu-trastuzumab. This is a radioactive tracer that was developed at MSKCC to target HER2 protein on cancer cells. A radioactive tracer is a small amount of radioactive dye that follows something else that is not radioactive In this study the study agent, 64Cu-trastuzumab, is the tracer and what's being followed is trastuzumab (Herceptin™). By giving you this tracer after you have treatment with trastuzumab (Herceptin™), we will be able to use PET scans to show us which parts of your body and tumor sites the Herceptin goes to. This will help us to understand better how Herceptin works in the body to fight cancer.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at MSKCC
* Age ≥18 years
* Patients with HER2+ metastatic breast cancer (either 3+ by immunohistochemistry or with evidence of gene amplification (>2.0) by fluorescence in situ hybridization (FISH))
* Measurable or evaluable disease
* Currently taking or about to commence treatment with trastuzumab at a dosing schedule of 2 mg/kg weekly or 6 mg/kg every three weeks, as per standard of care
* Karnofsky Performance Score ≥ 60
* Signed informed consent

Exclusion Criteria:

* Previous Grade 3 or higher allergic reaction to trastuzumab that resulted in discontinuation of trastuzumab therapy
* Claustrophobia/pain leading to inability to lie still for the duration of the scanning procedure.
* Pregnancy Test to be performed on female patients of childbearing potential within 24hrs before administration of radioactive material.
* Inability to provide written informed consent.
* Patients with liver metastases as the only site of distant disease
* Patients with known sensitivity or contraindication to Herceptin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
test safety & feas of (PET) imaging w radiolabeled 64Cu-trastuzumab to determine dosimetry & biodistribution of trastuzumab, using a radiotracer dilution technique w copper-64 labeled trastuzumab | conclusion of study

SECONDARY OUTCOMES:
to determine reproducibility of the measurement of the Standardized Uptake Value (SUV) in normal organs and tumors in a sub-cohort of 8 patients who will undergo two injections of the tracer. | conclusion of study
to determine the pharmacokinetic profile of the 64Cu-trastuzumab radiotracer. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Carrasquillo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org